CLINICAL TRIAL: NCT01219023
Title: Treatment of Palmar Plantar Erythrodysesthesia (PPE) With Topical Sildenafil
Acronym: JADE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00021480
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Hand Foot Syndrome; Palmar Plantar Erythrodysesthesia
Keywords: Hand foot syndrome; Palmar Plantar Erythrodysesthesia; chemotherapy; Sunitinib; Capecitebine; Sildenafil
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sildenafil citrate — Subjects will be given 2 types of topical creams, one containing 1% sildenafil and one containing placebo control. Subjects will be randomized to apply sildenafil cream to either the right or left hand/foot; placebo cream will be applied to the opposite hand/foot. The cream will be supplied to subjects with proper labeling to indicate right and left application assignment. Cream will be applied to each affected hand/foot two times per day.
  Other Names: Viagra

SUMMARY:
Hand-foot syndrome (HFS), also known as palmar-plantar erythrodysethesia (PPE), occurs in a 25%-50% of patients treated with several commonly used anti-cancer drugs including capecitabine and sunitinib. These drugs are known to improve survival in many cancers, including cancers of the colon, stomach, liver, breast, kidney, and GI stromal tumors (GIST). Worldwide, over 400,000 patients per year are treated with one of these agents. HFS involves skin changes, such as swelling, peeling, and blistering of the palms and soles, which is often painful and debilitating. As a result, HFS-related symptoms can frequently lead to dose reduction and/or discontinuation of otherwise effective anti-cancer treatment. There is no treatment for HFS other than dose reduction or stopping treatment. This proposal could quickly lead to treatments to prevent and/or treat HFS and help patients avoid debilitating side effects while continuing otherwise effective treatments for their cancer.

DETAILED DESCRIPTION:
The primary objective is to evaluate whether topical sildenafil reduces the severity of hand foot syndrome or palmar plantar erythrodysesthesia (PPE) associated with sunitinib and capecitabine. The secondary objective is to describe any toxicities associated with topical sildenafil.

This is a randomized, double blind, placebo-controlled pilot study of topical sildenafil for patients with grade 1-3 hand foot syndrome related to chemotherapeutic agents.

Approximately 20 evaluable patients with grade 1-3 PPE will be treated with topical sildenafil:

* 10 patients with PPE related to sunitinib
* 10 patients with PPE related to capecitabine

Once eligibility and screening criteria are met, subjects will be given 2 types of topical cream, one containing 1% sildenafil citrate and one containing placebo control. Subjects will be randomized to apply sildenafil citrate cream to either the right or left hand/foot; placebo cream will be applied to the opposite hand/ foot.

Clinical history, physical examination and photography of the hands and feet will be performed every two weeks for the first 2 months for patients on sunitinib and then every 4-6 weeks thereafter. For patients on capecitabine (which is given on an every 3 week schedule), these evaluations will be done every 3 weeks. Additional visits may be performed if clinically indicated.

If PPE resolves, less frequent administration and lower doses will be permitted to maintain responses. For consistency, patients may first reduce treatment to twice per day at the dose at which the PPE resolved. If this dosing schedule is effective then lower concentrations, e.g. 0.5%, may be used.

Patient cream assignment will be un-blinded at the 8 or 9 week time period (depending on the chemotherapy). However, patients with a 2 grade improvement in PPE in one hand versus the other (e.g. grade 3 improves to grade 1, or grade 2 improves to grade 0) that is maintained for at least 2 weeks, will be eligible for early un-blinding and treatment with active sildenafil for both hands and both feet.

Patients may receive topical sildenafil for up to 6 months on study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for the study:

1. Receiving capecitabine or sunitinib as part of routine standard care.
2. CTCAE version 4.0, grade 1-3 PPE.
3. Adults age ≥ 18
4. Karnofsky (KPS) performance status of ≥70%
5. Adequate organ and marrow function as defined below:

   1. - ANC > 1000/mL
   2. - Platelets > 75,000/mL
   3. - Total bilirubin < 1.5 x UNL
   4. - AST(SGOT)/ALT(SGPT) < 5 x UNL
   5. - Creatinine Cr Cl est > 40 mL/min (by Cockcroft-Gault)
6. Not pregnant or lactating.
7. Use of adequate birth control with female partners of male subjects agreeing to use a medically acceptable form of birth control: (1) surgical sterilization, (2) approved hormonal contraceptives (such as birth control pills or Depo-Provera), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, (4) an intrauterine device (IUD) or (5) post menopausal. Abstinence is not considered acceptable birth control. Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Subjects meeting any of the following criteria are ineligible for study entry:

1. Currently participating in a clinical trial.
2. History of hypersensitivity or intolerance to sildenafil or other related products tadalafil (Cialis™), vardenafil (Levitra™) or poloxamer vehicle.
3. Currently taking oral sildenafil or other related products tadalafil (Cialis™), vardenafil (Levitra™).
4. Currently taking other treatment for PPE other than standard emollients.
5. Using organic nitrates, either regularly and/or intermittently, in any form.
6. History of myocardial infarction, stroke, or life-threatening arrhythmia within the last 6 months.
7. Resting hypotension (BP <90/50 mmHg) or hypertension (BP >170/110 mmHg). Those subjects on alpha-blocker or anti-hypertensive therapy must be hemodynamically stable for at least two weeks before day 1 of study drug.
8. Cardiac failure or coronary artery disease causing unstable angina.
9. Known retinitis pigmentosa (a minority of these patients have genetic disorders of retinal phosphodiesterases).
10. Concomitant use of strong cytochrome P450 3A4 inducers or inhibitors (Ex: ketoconazole, itraconazole, erythromycin, saquinavir).
11. Other acute or chronic inflammatory conditions or infections of the hands or feet that would complicate safety, application of topical creams, or study endpoints.
12. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
13. Pregnant or breast-feeding and/or lactating.
14. Inability or unwillingness to comply with protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Grade of hand foot syndrome over time as measured by NCI CTC version 4.0 PPE syndrome criteria | Every 2 weeks (sunitinib arm); Every 3 weeks (capecitabine arm)
  Grading of PPE by NCI CTC criteria occurs every 2 weeks for subjects in the sunitinib arm for 1st 8 weeks (and as clinically indicated). Grading of PPE by NCI CTC criteria occurs every 3 weeks for subjects in the capeccitabine arm for the 1st 9 weeks (and as clinically indicated)
Assessment of patient reported pain, at rest and when making a fist, using a 1-10 score. | twice daily
  Assessment of patient reported pain, at rest and when making a fist, using a 1-10 score, is collected on a diary card that subjects fill out twice daily.
Assessment of severity of erythema and desquamation or blistering as measured on 0-4 score from photographs. | Every 2 weeks (sunitinib arm); Every 3 weeks (capecitabine arm)
  Assessment of severity of erythema and desquamation or blistering as measured on 0-4 score from photographs of hands and/or feet taken every two weeks (for subjects in sunitinib arm) or every 3 weeks (for subjects in capecitabine arm).

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States